CLINICAL TRIAL: NCT04452578
Title: Pilot Investigation Using HCV Positive Heart Grafts in HCV Negative or Previously Successfully Treated Recipients
Brief Title: Hepatitis C Virus (HVC) Positive Heart Grafts in HCV Negative Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5190371
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure
Keywords: HCV
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Recipient of HCV positive heart graft (Experimental): A single center, open-label, pilot study examining 10 adult HCV negative heart transplant subjects who will receive an HCV infected graft. Target start date for antiviral therapy will be within 3 months after heart transplantation.
  Interventions: Procedure: Procedure: Heart Transplantation

INTERVENTIONS:
Procedure: Procedure: Heart Transplantation — A HCV negative or previously successfully treated recipient who recieves a HCV positive graft will be monitored. Patients who recieve an HCV graft will be treated for HCV according to accepted protocols.

SUMMARY:
To provide proof-of-concept data on the efficacy/safety of transplanting HCV positive donor grafts in HCV negative heart recipients who are currently listed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 and older
* Active on the transplant list
* Donor organ with Antibody and NAT (nucleic acid test) positive for HCV
* HCV negative recipient; this includes patients who never had HCV and those with HCV previously eradicated with antiviral therapy. The latter is defined as those with undetectable HCV viral load at least 3 months since stopping therapy.
* Willing and able to provide written informed consent or for those subjects where hepatic encephalopathy affects their ability to provide initial or ongoing consent, has an appropriate and legally-authorized representative willing and able to provide consent on behalf of the subject
* Patients listed for multiple organ transplant (heart and kidney or heart and liver) can be included based on agreement of non-cardiac organ transplant team

Exclusion Criteria:

* Participants co-infected with HIV
* Donor previously treated with an NS5a containing regimen (if treatment history of donor known)
* Known allergies or hypersensitivity to DAA or ribavarin
* Pregnancy and/or actively breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Patient Survival Rate | 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Transplant Institute, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No